CLINICAL TRIAL: NCT02614768
Title: Standardized Evaluation of Subcutaneous Glucose Monitoring Systems Under Routine Environmental Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SPIDIMAN_01
Record Dates: First submitted 2015-11-24; First posted 2015-11-25 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Glucose Monitoring System
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glucose Sensor (Experimental): Continuous subcutaneous glucose monitoring using four different CGM systems in parallel will be performed throughout the study. Insulin therapy will be performed by the subjects themselves, as under daily life conditions. For the hypoglycaemia experiment an increased insulin bolus will be administered with meals (180% of the subject's calculated mealtime dose).
  Interventions: Device: Glucose Sensor

INTERVENTIONS:
Device: Glucose Sensor — The investigational intervention is CGM monitoring using four different CGM systems. Three of the four CGM devices which are used will be CGM systems which have received conformité européenne (CE) certification (Dexcom G4 Platinum, Medtronic MiniMed 640G system, Abbott FreeStyle Libre Flash). The SPIDIMAN sensor will be used for the first time in human subjects, does not yet have received CE certification and will be given an identifying label in addition to being labelled "for investigative use only".

SUMMARY:
The purpose of this study is to assess accuracy and reliability of the SPIDIMAN continuous glucose monitoring (CGM) sensor system with regard to values as measured by Super GL and compare these results with similar evaluations of the Medtronic MiniMed 640G system, the Abbott FreeStyle Libre Flash Sensor and the DexCom G4 Platinum Sensor in patients with type 1 Diabetes.

DETAILED DESCRIPTION:
The study is a single-center open-label study in patients with type 1 diabetes treated with continuous subcutaneous insulin infusion (CSII) or multiple daily injections (MDI) therapy. The study will include a total of 12 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained after being advised of the nature of the study
* Male or female aged ≥18 years
* Type 1 diabetes for at least 6 months according to the World Health Organization (WHO) definition
* Treatment with multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII) for at least 3 months
* Body Mass Index (BMI) < 35 kg/m²
* Willing and able to wear 5 CGM devices for the duration of the study and undergo all study procedures.
* HbA1c ≤ 86 mmol/mol

Exclusion Criteria:

* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the subject
* Female of childbearing potential who is pregnant, breast-feeding or intend to become pregnant or is not using adequate contraceptive methods
* Any mental condition rendering the subject incapable of giving his consent
* Subject is using a medication that significantly impacts glucose metabolism (oral steroids) except if stable for at least the last three months and expected to remain stable for the study duration
* Subject may not use acetaminophen (paracetamol) while participating in the study
* Has severe medical or psychological condition(s) or chronic conditions/infections that in the opinion of the Investigator would compromise the subject's safety or successful participation in the study.
* Subject is actively enrolled in another clinical trial
* Known adrenal gland problem, pancreatic tumour, or insulinoma
* Inability of the subject to comply with all study procedures
* Inability of the subject to understand the patient information.
* Subject donated blood in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Mader, Prof. Dr., Principal Investigator — Medical University of Graz

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glucose Sensor
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Glucose Sensor
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Europe | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Test-to-Reference Measurement Pairs With an Absolute Relative Difference (ARD) ≤15%
Description: The primary outcome measure was overall sensor accuracy determined using ISO 15197:2013, which is percentage (%) of sensor values that are within ±0.8 mmol/L of the reference value at glucose concentrations <5.6 mmol/L and within ±15% at glucose concentrations ≥5.6 mmol/L. The sensor values were obtained using three different glucose monitoring systems, i.e. Abbott, Dexcom and Medtronic, in patients with T1D over a 12-hour period in standardized conditions. The reference values were obtained by analysis of venous plasma glucose samples.
Time Frame: 36 hours
Measure: Number; unit: Percentage of sensor values
Arm/Group | Glucose Sensor
Number analyzed (Participants) | 12
Percentage of sensor values
  Abbot | 73.2
  Dexcom | 56.1
  Medtronic | 52.0

ADVERSE EVENTS:
Arm/Group | Glucose Sensor
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glucose Sensor (N=12)
Superficial excoriation (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes